CLINICAL TRIAL: NCT05048706
Title: Comparative Effectiveness of the Super Pulse Thulium Fiber Laser (SP TLF) for Laser Lithotripsy of Urinary Calculi
Brief Title: SP TLF Versus Ho:YAG Laser
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00005201
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Urinary Calculi
MeSH Terms: conditions — Urinary Calculi | interventions — Lithotripsy, Laser

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Super Pulse Thulium fiber Laser
  Interventions: Device: Laser lithotripsy (SP TLF)
- Holmium: Yttrium-Aluminium-Garnet Laser
  Interventions: Device: Laser lithotripsy (Ho:YAG)

INTERVENTIONS:
Device: Laser lithotripsy (SP TLF) — Laser lithotripsy of urinary calculi using the Super Pulse Thulium fiber laser (SP TLF)
  Groups: Super Pulse Thulium fiber Laser
Device: Laser lithotripsy (Ho:YAG) — Laser lithotripsy of urinary calculi using the standard Holmium: Yttrium-Aluminium-Garnet (Ho:YAG) laser.
  Groups: Holmium: Yttrium-Aluminium-Garnet Laser

SUMMARY:
The investigators aim to compare the performance of the Super Pulse Thulium fiber laser (SP TFL) with that of the standard Holmium: Yttrium-Aluminium-Garnet (Ho:YAG) laser. The investigators hypothesize that the electronically-modulated laser diodes, of the TFL offers the most comprehensive and flexible range of laser parameters among laser lithotripters leading to more efficient (4 times more) and effective stone dusting resulting in production of finer dust particles obviating the need for postoperative ureteric stenting which remains a major source of patient discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Patient is scheduled to undergo mini-PCNL and/or RIRS surgery at the University of Rochester Medical Center for the management of upper urinary tract calculi (i.e. kidney and proximal ureter)
* Stones located in the kidney and proximal ureter
* Stones measuring 10-30mm
* Ability to give informed consent
* Any racial or ethnic origin
* Age 18 years and older

Exclusion Criteria:

* Active kidney infection
* Patients with prior stenting
* Pregnant patients
* Patients with solitary kidney
* Patients with ureteral tumor or stricture
* Inability to give informed consent
* Not age 18 and older

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects eligible for this study will be identified via eRecord in the Urology Department (routine access) of patients who were diagnosed with upper urinary tract calculi who underwent surgery utilizing either high powered Ho:YAG or TL-SPL lasers.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
To determine the efficiency of SP TFL in dusting stones | 6 months
  We plan to assess the direct impact of SP TFL to efficiently dust 10-30mm stones in the upper urinary tract . Metrics include time needed to ablate the stone i.e. ablation speed (stone volume mm3/sec)
Mean ablation energy needed to ablate stone volume | 6 months
  We plan to assess the direct impact of SP TFL to effectively dust 10-30mm stones in the upper urinary tract . Metrics include ablation energy needed to ablate the stone volume (Stone volume mm3/Joules)

SECONDARY OUTCOMES:
Number of stones cleared. | 9 months
  We plan to assess the direct impact of SP TFL to produce finer quality dust following disregarding of 10-30mm stones in the upper urinary tract that can spontaneously pass without the need for stenting . Metrics will be stone clearance on postoperative CT scans
Number of participants reporting complications. | 9 months
  We plan to assess the direct impact of SP TFL to safely dust 10-30mm stones in the upper urinary tract . Metrics collected will include review of medical record for the presence of complications (e.g. infection, sepsis, obstruction etc.) for 3 months postoperative related to laser lithotripsy.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Ghazi, MD, Principal Investigator — Associate Professor
Locations (2):
- United States (2):
  - University of Rochester Medical Center, Rochester, New York
  - University of Rochester, Rochester, New York

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers.